CLINICAL TRIAL: NCT02278419
Title: A Phase 2a, Partly Randomized, Open-label Trial to Investigate the Efficacy and Safety of an 8 or 12-Week Treatment Regimen of Simeprevir in Combination With Sofosbuvir in Treatment-Naive and Experienced Subjects With Chronic Genotype 4 Hepatitis C Infection
Brief Title: An Efficacy and Safety Study of a 8 or 12-Week Treatment Regimen of Simeprevir in Combination With Sofosbuvir in Treatment-Naive and Experienced Participants With Chronic Genotype 4 Hepatitis C Virus Infection
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Janssen-Cilag International NV (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CR104970; TMC435HPC2014 (Other: Janssen-Cilag International NV)
Record Dates: First submitted 2014-10-28; First posted 2014-10-30 (Estimated); Last update posted 2016-10-14 (Estimated); Status verified 2016-09

CONDITIONS: Hepatitis C
Keywords: Hepatitis C; Simeprevir; Sofosbuvir; Healthy
MeSH Terms: conditions — Hepatitis C | interventions — Simeprevir; Sofosbuvir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Group A1 (Experimental): Participants without cirrhosis will receive simeprevir 150 milligram (mg) capsule along with sofosbuvir 400 mg tablet, orally, once daily for 8 weeks.
  Interventions: Drug: Simeprevir; Drug: Sofosbuvir
- Group A2 (Experimental): Participants without cirrhosis will receive simeprevir 150 mg capsule along with sofosbuvir 400 mg tablet, orally, once daily for 12 weeks.
  Interventions: Drug: Simeprevir; Drug: Sofosbuvir
- Group B (Experimental): Participants with cirrhosis will receive simeprevir 150 mg capsule along with sofosbuvir 400 mg tablet, orally, once daily for 12 weeks.
  Interventions: Drug: Simeprevir; Drug: Sofosbuvir

INTERVENTIONS:
Drug: Simeprevir — Simeprevir 150 mg capsule orally, once daily for 8 weeks in Group A1, 12 weeks in Group A2 and Group B.
Drug: Sofosbuvir — Sofosbuvir 400 mg tablet orally, once daily for 8 weeks in Group A1, 12 weeks in Group A2 and Group B.

SUMMARY:
The purpose of this study is to evaluate the efficacy of simeprevir in combination with sofosbuvir for 8 or 12 weeks versus a historical control, with respect to the percentage of participants with sustained virologic response at 12 weeks after end of treatment (SVR12) in the overall population.

DETAILED DESCRIPTION:
This is a partly randomized, open-label (identity of study drug will be known to volunteer and study staff), multicenter (when more than one hospital or medical school team work on a medical research study) study. The study will consist of a screening period of up to 4 weeks, an open-label treatment period of 8 weeks or 12 weeks, and a post-treatment follow-up period until 24 weeks after end of treatment (EOT). Participants without cirrhosis will be assigned to Group A wherein half of the participants will receive 8 week treatment in Group A1 and remaining participants will receive 12 week treatment in Group A2. Participants with cirrhosis, will be assigned to Group B to receive simeprevir in combination with sofosbuvir for 12 weeks. The duration of participation for each participant, including the screening period, will be approximately 36 or 40 weeks for 8 or 12 week treatment, respectively. Efficacy will be primarily assessed by percentage of participants with SVR12. Participants' safety will be evaluated throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Participant must have hepatitis C virus (HCV) genotype 4 infection (confirmed at screening)
* Participant must have HCV ribonucleic acid (RNA) greater than (>) 10,000 international unit per milliliter (IU/mL) at screening
* In participants with cirrhosis, a documented hepatic imaging procedure (ultrasound, computed tomography [CT] scan, or magnetic resonance imaging [MRI]) within 6 months before baseline (Day 1) to exclude hepatocellular carcinoma is required
* A woman of childbearing potential must have a negative serum (beta human chorionic gonadotropin at screening and a negative urine pregnancy test on Day 1 before first dose of study drug
* Females of childbearing potential or males with a female partner of childbearing potential must agree to use 2 highly effective contraceptive methods (one of which is a barrier method; eg, condom or diaphragm) from Day 1 (baseline) and continue until 30 days after the end of treatment (EOT) (or longer if dictated by local regulations), or not be heterosexually active, or be a vasectomized male subject or a female subject with a vasectomized partner, or be a female (subject or partner of male subject) of non-childbearing potential (ie, postmenopausal for at least 2 years or surgically sterile)

Exclusion Criteria:

* Participant has evidence of clinical hepatic decompensation (history or current evidence of ascites, bleeding varices, or hepatic encephalopathy)
* Participant has any liver disease of non-HCV etiology. This includes, but is not limited to, acute hepatitis A, drug- or alcohol-related liver disease, autoimmune hepatitis, hemochromatosis, Wilson's disease, alpha-1 antitrypsin deficiency, non-alcoholic steatohepatitis, primary biliary cirrhosis, or any other non-HCV liver disease considered clinically significant by the investigator
* Participant is infected/co-infected with non-genotype 4 HCV
* Participant has any other active clinically significant disease or clinically significant findings during screening of medical history, physical examination, laboratory testing or electrocardiogram (ECG) recordings that, in the investigator's opinion, would compromise the participant's safety or could interfere with the participant participating in and completing the study
* Participant has history of malignancy within 5 years of the screening visit (exceptions: skin carcinomas, carcinoma in situ of the cervix, or malignancy that in the opinion of the investigator is considered cured with minimal risk of recurrence)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2014-12; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants With Sustained Virologic Response at Week 12 After End of Treatment (SVR12) | 12 weeks after end of treatment (EOT) (EOT; Week 8 for Group A1, Week 12 for Group A2 and Group B)
  SVR12 is defined as hepatitis C virus (HCV) ribonucleic acid (RNA) less than (<) lower limit of quantification (LLOQ; 15 international unit per milliliter [IU/mL]), detectable or undetectable at 12 weeks after EOT.

SECONDARY OUTCOMES:
Percentage of Participants With Sustained Virologic Response at Week 4 After End of Treatment (SVR4) | 4 weeks after EOT (EOT; Week 8 for Group A1, Week 12 for Group A2 and Group B)
  SVR4 is defined as HCV RNA <LLOQ;15 IU/mL, at 4 weeks after EOT.
Percentage of Participants With Sustained Virologic Response at Week 24 After End of Treatment (SVR24) | 24 weeks after EOT (EOT; Week 8 for Group A1, Week 12 for Group A2 and Group B)
  SVR24 is defined as HCV RNA <LLOQ;15 IU/mL, at 24 weeks after EOT.
Percentage of Participants With on-treatment Failure | EOT (EOT; Week 8 for Group A1, Week 12 for Group A2 and Group B)
  Participants will be considered on-treatment failures if they have (confirmed) detectable HCV RNA, that is <LLOQ;15 IU/mL, detectable or greater than or equal to (>=) LLOQ at EOT.
Percentage of Participants With Viral Relapse | EOT (Week 8 for Group A1, Week 12 for Group A2 and Group B), Weeks 4, 12 and 24 after end of treatment
  Participants will be considered to have viral relapse if they do not achieve SVR at Week 4, 12 and 24 after EOT and meet the following conditions 1) HCV RNA <LLOQ;15 IU/mL, undetectable at EOT, 2) HCV RNA >=LLOQ;15 IU/mL during the follow-up period.
Percentage of Participants With On-treatment Response | Week 1, 2, 4, 8 and EOT for all groups, Week 12 for Group A2 and Group B
  On-treatment virologic response is defined as the change from baseline in log10 hepatitis C virus ribonucleic acid.
Percentage of Participants With Viral Breakthrough | Week 1 up to Week 8 in Group A1, Week 1 up to Week 12 in Group A2 and Group B
  Viral breakthrough is defined as confirmed >1.0 log10 increase in HCV RNA from nadir or confirmed HCV RNA >100 IU/mL in participants who had previously achieved HCV RNA <LLOQ; 15 IU/mL.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen-Cilag International NV Clinical Trial, Study Director — Janssen-Cilag International NV
Locations (2):
- Egypt (2):
  - Cairo
  - Menoufiya

REFERENCES:
- [Derived] El Raziky M, Gamil M, Ashour MK, Sameea EA, Doss W, Hamada Y, Van Dooren G, DeMasi R, Keim S, Lonjon-Domanec I, Hammad R, Hashim MS, Hassany M, Waked I. Simeprevir plus sofosbuvir for eight or 12 weeks in treatment-naive and treatment-experienced hepatitis C virus genotype 4 patients with or without cirrhosis. J Viral Hepat. 2017 Feb;24(2):102-110. doi: 10.1111/jvh.12625. Epub 2016 Oct 27. PMID 27790789
- See also: A Phase2a,Partly Randomized,Open-label Trial to Investigate the Efficacy and Safety of an 8 or 12 Week Treatment Regimen of Simeprevir in CombinationWith Sofosbuvir in Treatment-Naïve and Experienced Subjects With Chronic Genotype 4 HepatitisC Infection — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_7051&studyid=7813&filename=CR104970_CSR.pdf